CLINICAL TRIAL: NCT05688618
Title: Effect of the Administration of a Symbiotic (E. Faecium and Agave Inulin) on Mild Cognitive Impairment in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anahuac University (Other)
Responsible Party: Principal Investigator, Jose Juan Antonio Ibarra Arias, Responsable, Anahuac University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CEI-004-20160729
Record Dates: First submitted 2022-08-19; First posted 2023-01-18 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator)
  Interventions: Dietary Supplement: Enteroccocus Facieum and Agave Inulin
- Control group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Enteroccocus Facieum and Agave Inulin — A pack of symbiotic powder with 1 gram of e. facieum and 8g of agave inulin will be administered daily for 8 weeks
  Arms: Experimental group
Other: Placebo — A pack of unsweetened almond powder milk will be administered daily for 8 weeks
  Arms: Control group

SUMMARY:
Cognitive impairment is one of the fastest growing diseases in the last decades, given the significant increase in senior citizen population in Mexico and the world.

Several studies have discussed the gut-microbiota-brain axis. It has been demonstrated that a balanced gut microbiota, prevents an increase in pro-inflammatory cytokines that affect specific brain areas; having an important impact at the cortical level of the hippocampus which translates to diminished cognitive function and the start of cognitive impairment symptoms.

After multiple studies on the effect of the administration of symbiotics in animal models in cognition and memory, there have been positive results, observing improvement in cognition and decrement in inflammatory cytokines at hippocampus level.

DETAILED DESCRIPTION:
Cognitive impairment is one of the fastest growing diseases in the last decades, given the significant increase in senior citizen population in Mexico and the world.

Cognitive impairment is the loss of cognitive functions, in the abscence of other pathologies that may be the cause of the memory loss. It is well known that this pathology can progress to more severe states reaching irreversible dementia such as Alzheimer in a short period of approximately 5 years from the onset of the disease.

Given the rapid increase in incidence of cognitive impairment, there have been several studies on the management of symptoms and on the natural course of the disease.

Several studies have discussed the gut-microbiota-brain axis. It has been demonstrated that a balanced gut microbiota, prevents an increase in pro-inflammatory cytokines that affect specific brain areas; having an important impact at the cortical level of the hippocampus which translates to diminished cognitive function and the start of cognitive impairment symptoms.

After multiple studies on the effect of the administration of symbiotics in animal models in cognition and memory, there have been positive results, observing improvement in cognition and decrement in inflammatory cytokines at hippocampus level.

The objective of this study is to evaluate the effect of the symbiotic on the cognitive process in senior adults.

To achieve this a clinical trial will be held in a senior citizen population who will be administered a symbiotic compound (enterococcus faecium and inulin) for 8 weeks and evaluated for cognitive functions using Mini-mental state examination, rey-osterrieth complex, and a validated tool (AeRAC).

The variables will be expressed as mean ± standard deviation, depending on the type of distribution of the data. It will be used paired T Student for homogenous data in an intragroup comparison or Wilcoxon test for heterogenous data. For intergroup comparison it will be used independent T Student for homogenous data and U Mann Whitney for dependent group in heterogenous data. Data analysis will be carried out using the latest version of GraphPad Prism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild cognitive impairment
* Patients who sign the informed consent

Exclusion Criteria:

* Patients who do not have mild cognitive impairment
* Patients with advanced cognitive impairment such as Alzheimers disease
* Patients with comorbidities that influence the cognitive functions such as diabetes mellitus, cerebral ischemia or previous brain trauma
* Patients who do not sign the informed consent

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment | 8 weeks
  Change in Score for Mini mental state examination
Cognitive impairment | 8 weeks
  Change in Score for Rey-Osterrieth complex figure
Cognitive impairment | 8 weeks
  Change in Score for AeRAC (Instrumento de expectativas de autoeficacia)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital ABC Santa Fe, Mexico City, Mexico

REFERENCES:
- [Background] Borras Blasco C, Vina Ribes J. [Neurophysiology and ageing. Definition and pathophysiological foundations of cognitive impairment]. Rev Esp Geriatr Gerontol. 2016 Jun;51 Suppl 1:3-6. doi: 10.1016/S0211-139X(16)30136-6. Spanish. PMID 27719970
- [Background] Benavides-Caro, C. Deterioro cognitivo en el adulto mayor. Medigraphic, (2017). 40(2).
- [Background] Romo-Araiza A, Gutierrez-Salmean G, Galvan EJ, Hernandez-Frausto M, Herrera-Lopez G, Romo-Parra H, Garcia-Contreras V, Fernandez-Presas AM, Jasso-Chavez R, Borlongan CV, Ibarra A. Probiotics and Prebiotics as a Therapeutic Strategy to Improve Memory in a Model of Middle-Aged Rats. Front Aging Neurosci. 2018 Dec 18;10:416. doi: 10.3389/fnagi.2018.00416. eCollection 2018. PMID 30618722
- [Background] Landefeld, C. Current geriatric diagnosis & treatment. New York: McGraw-Hill Professional. (2004).
- [Background] Lin JS, O'Connor E, Rossom RC, Perdue LA, Eckstrom E. Screening for cognitive impairment in older adults: A systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2013 Nov 5;159(9):601-12. doi: 10.7326/0003-4819-159-9-201311050-00730. PMID 24145578
- [Background] Grammas P. Neurovascular dysfunction, inflammation and endothelial activation: implications for the pathogenesis of Alzheimer's disease. J Neuroinflammation. 2011 Mar 25;8:26. doi: 10.1186/1742-2094-8-26. PMID 21439035
- [Background] Ticinesi A, Tana C, Nouvenne A, Prati B, Lauretani F, Meschi T. Gut microbiota, cognitive frailty and dementia in older individuals: a systematic review. Clin Interv Aging. 2018 Aug 29;13:1497-1511. doi: 10.2147/CIA.S139163. eCollection 2018. PMID 30214170
- [Background] Novotny M, Klimova B, Valis M. Microbiome and Cognitive Impairment: Can Any Diets Influence Learning Processes in a Positive Way? Front Aging Neurosci. 2019 Jun 28;11:170. doi: 10.3389/fnagi.2019.00170. eCollection 2019. PMID 31316375
- [Background] Dalile, B., Verbeke, K., Van Oudenhove, L. and Vervliet, B. Nourishing the gut microbiota: The potential of prebiotics in microbiota-gut-brain axis research. Behavioral and Brain Sciences, (2019). 42.
- [Background] Quigley EM. Prebiotics and probiotics; modifying and mining the microbiota. Pharmacol Res. 2010 Mar;61(3):213-8. doi: 10.1016/j.phrs.2010.01.004. Epub 2010 Jan 18. PMID 20080184
- [Background] Olveira G, Gonzalez-Molero I. An update on probiotics, prebiotics and symbiotics in clinical nutrition. Endocrinol Nutr. 2016 Nov;63(9):482-494. doi: 10.1016/j.endonu.2016.07.006. Epub 2016 Sep 12. English, Spanish. PMID 27633133
- [Background] Bautista Justo, M.; García Oropeza, L.; Salcedo Hernández, R.; Parra Negrete, L. A. Azúcares en agaves (agave tequilana Weber) cultivados en el estado de guanajuato Acta Universitaria, vol. 11, núm. 1, abril, 2001, pp. 33-38
- [Background] Louzada ER, Ribeiro SML. Synbiotic supplementation, systemic inflammation, and symptoms of brain disorders in elders: A secondary study from a randomized clinical trial. Nutr Neurosci. 2020 Feb;23(2):93-100. doi: 10.1080/1028415X.2018.1477349. Epub 2018 May 23. PMID 29788823
- [Background] Ginsberg TB, Powell L, Emrani S, Wasserman V, Higgins S, Chopra A, Cavalieri TA, Libon DJ. Instrumental Activities of Daily Living, Neuropsychiatric Symptoms, and Neuropsychological Impairment in Mild Cognitive Impairment. J Am Osteopath Assoc. 2019 Feb 1;119(2):96-101. doi: 10.7556/jaoa.2019.015. PMID 30688355
- [Background] Pita Fernández, S., Pértega Díaz, S., Unidad de Epidemiología Clínica y Bioestadística. Complexo Hospitalario Universitario de A Coruña (España) CAD ATEN PRIMARIA 2001; 8: 191-195
- [Background] Hanchi H, Mottawea W, Sebei K, Hammami R. The Genus Enterococcus: Between Probiotic Potential and Safety Concerns-An Update. Front Microbiol. 2018 Aug 3;9:1791. doi: 10.3389/fmicb.2018.01791. eCollection 2018. PMID 30123208
- [Background] Aguirre Leuke, Probióticos, prebióticos y simbióticos. El farmacéitico. 2017;542 pp. 25- 24
- [Background] Shi Y, Zhai M, Li J, Li B. Evaluation of safety and probiotic properties of a strain of Enterococcus faecium isolated from chicken bile. J Food Sci Technol. 2020 Feb;57(2):578-587. doi: 10.1007/s13197-019-04089-7. Epub 2019 Sep 11. PMID 32116367
- [Background] Rogers GB, Keating DJ, Young RL, Wong ML, Licinio J, Wesselingh S. From gut dysbiosis to altered brain function and mental illness: mechanisms and pathways. Mol Psychiatry. 2016 Jun;21(6):738-48. doi: 10.1038/mp.2016.50. Epub 2016 Apr 19. PMID 27090305
- See also: Related Info — https://www.who.int/es/news-room/fact-sheets/detail/dementia
- See also: Related Info — https://doi.org/10.3389/fmicb.2018.01791
- See also: Related Info — http://www.conapo.gob.mx/work/models/CONAPO/Resource/1529/2/images/DocumentoMetodologicoProyecciones2010_2050.pdf
- Available data/document: Study Protocol — https://drive.google.com/drive/u/0/folders/1JG22lkEchQULxW79ktlsVcM5uGNB4iVh